CLINICAL TRIAL: NCT06991010
Title: One-arm, Prospective, Clinical Use Study of the Suction-Activated Patent Hemostasis (SAPH) Device After a Transradial Procedure
Brief Title: Clinical Use Study of SAPH Device for Patent Hemostasis After a Transradial Procedure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Transradial Technologies, LLC (Industry)
Collaborators: RARAS CRO (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT012025
Record Dates: First submitted 2025-04-25; First posted 2025-05-25 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hemostasis of Arterial Punctures
Keywords: Artery clamp; Transradial access; Radial artery patency; Radial artery hemostasis

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, nonrandomized, single-cohort, interventional clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- SAPH Device (Experimental): All patients who have the SAPH device used to achieve hemostasis
  Interventions: Device: Suction-Activated Patent Hemostasis (SAPH) Device

INTERVENTIONS:
Device: Suction-Activated Patent Hemostasis (SAPH) Device — A compression device intended to achieve patient hemostasis of the radial artery

SUMMARY:
This is a prospective, multicenter study intended to provide supportive clinical information on the use of the SAPH device to achieve radial artery patent hemostasis after a transradial procedure.

DETAILED DESCRIPTION:
This is a prospective, multicenter, nonrandomized, single-cohort, interventional clinical study intended to provide supportive clinical information to the nonclinical characterization and performance data required for demonstration of substantial equivalence to marketed devices. The study will assess clinical use elements such as ease of use, patient comfort, as well as safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 21 years or older.
2. Patient is scheduled to undergo a coronary or peripheral catheterization procedure requiring 5 or 6 Fr transradial sheath access (TRA) with planned same-day discharge
3. Patient has a Reverse Barbeau test result of Type A, B or C (patent radial artery)
4. Patient is able to understand informed consent language
5. Patient is willing and able to sign informed consent and adhere to the protocol requirements

Exclusion Criteria:

1. Patient had a prior ipsilateral TRA procedure
2. Patient has scleroderma, vasculitis, or Raynaud's syndrome (primary or secondary)
3. Patient has cellulitis overlying radial artery
4. Patient requires uninterrupted oral systemic anticoagulation
5. Patient has intolerance to standard anticoagulants used in TRA procedures
6. Patient has non-palpable radial pulse or Reverse Barbeau test Type D response
7. Patient is participating in another investigational study
8. Patient is a prisoner
9. Patient, in the principal investigator's opinion, would not be able to comply with protocol requirements including self-report of comfort and 30-day follow up
10. Patient is receiving glycoprotein IIb/IIIa inhibitors
11. Patients with allergy to medical adhesives

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
Efficacy Endpoint - Percent of subjects with radial artery hemostasis with patency at time of discharge | 60 minutes prior to same-day discharge or within 24 hours post-TRA procedure.
  Radial artery hemostasis with patency is defined as hemostasis over the arterial puncture site with palpable distal radial pulse or prominent digital arterial waveform signal by digital plethysmography with ulnar occlusion.
Safety Endpoints - 1) Percentage of subjects with radial artery patency 2) No major device-related access site-related complications prior to discharge | 60 minutes prior to same-day discharge or within 24 hours post-TRA procedure
  Patency is defined as prominent digital arterial waveform signal by digital plethysmography with ulnar artery occlusion.

CONTACTS AND LOCATIONS:
Overall Officials: Regulatory and Clinical Lead, PhD, Study Director — Transradial Technologies, LLC

IPD SHARING:
Plan to Share IPD: Undecided